CLINICAL TRIAL: NCT00420771
Title: A Randomized Controlled Pilot Trial of Gabapentin for the Treatment of Benzodiazepine Abuse in Methadone Maintenance Patients
Brief Title: Gabapentin Treatment of Benzodiazepine Abuse in Methadone Maintenance Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, John Mariani MD, research psychiatrist, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4906/#5998R; K23DA021209 (NIH)
Record Dates: First submitted 2007-01-08; First posted 2007-01-11 (Estimated); Results first posted 2018-07-12 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Benzodiazepine Dependence; Opioid Dependence
Keywords: Benzodiazepine; Gabapentin; Methadone
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gabapentin (Experimental): gabapentin treatment 1200 mg three times daily
  Interventions: Drug: Gabapentin
- Placebo (Placebo Comparator): Placebo condition received pills identical in appearance to experimental arm.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gabapentin — For the first week, one 400 mg Gabapentin capsule taken 3 times per day. For the second week, two 400 mg Gabapentin capsules taken 3 times per day. For the third week through the eighth week, three 400 mg Gabapentin capsules taken 3 times per day. For the ninth and last week, two 400 mg Gabapentin capsules taken 3 times per day for 3 days, then one 400 mg Gabapentin capsule taken 3 times per day for 4 days. Placebo study medication appears identical to active medication and is prescribed with an identical dosing schedule.
  Other Names: Neurontin
  Arms: Gabapentin
Drug: Placebo — placebo comparator appears identical to active medication and is prescribed with an identical dosing schedule with a maximum dose of 400mg taken three times per day
  Arms: Placebo

SUMMARY:
The aim of this project is to study the use of gabapentin in reducing benzodiazepine abuse in methadone maintenance patients. A second aim is to study the effects of gabapentin on craving, mood, anxiety, and sleep disturbance in methadone maintenance patients abusing benzodiazepines. The proposed protocol is a randomized, double-blind, placebo-controlled pilot outpatient trial of gabapentin in the treatment of benzodiazepine abuse in methadone maintenance patients. All subjects will receive weekly manual-guided psychotherapy directed at achieving abstinence and improving current functioning. The primary outcome measure, benzodiazepine use, will be assessed weekly by a combination of self-report (time line follow-back method) and urine toxicology. Associated psychological symptoms of craving, mood, anxiety, and sleep disturbance, will be assessed by a combination of clinician and self-rated instruments.

The investigators hypothesize that individuals receiving methadone maintenance treatment who are abusing (nonprescribed use) benzodiazepines have difficulty in reducing or discontinuing benzodiazepine use because of the significant anxiety, mood, and sleep disturbance symptoms that accompany reduction in use. Gabapentin, an anticonvulsant which has anxiolytic and sedating properties, may alleviate the symptoms associated with a reduction in benzodiazepine abuse and make the achievement of abstinence more likely when administered in the setting of an active psychotherapy condition.

DETAILED DESCRIPTION:
The investigators will recruit individuals with current benzodiazepine abuse or dependence, as defined by the DSM-IV, who are receiving methadone maintenance treatment at the Bridge Plaza Treatment and Rehabilitation Clinic. The initial step in recruitment for all patients will be a referral from a clinic counselor.

The investigators plan to enroll 86 participants into the study. Both males and females will be recruited. The distribution of benzodiazepine abuse in methadone maintenance populations with regard to race and gender is not well studied.The investigators expect the gender and racial distribution of subjects to reflect the demographic nature of the Bridge Plaza Treatment and Rehabilitation Clinic; which is approximately 33% Caucasian, 33% African-American, and 33% Hispanic; and 40% female. The investigators will make every effort to recruit minority patients in order to ensure the ability to generalize our findings to the overall treatment population.

All patients will begin medication at the start of the study. Subjects will take medication twice each day, once in the morning and once in the evening. All tablets (placebo and study medication) will be over-capsulated with riboflavin to measure compliance. The placebo group will have a dosing schedule that is identical to the gabapentin group (i.e., they will take the same number of pills each day). Medication will be dispensed weekly in individual vials identified by patient, with dosing instructions written on the outside of the vials. Patients in the placebo group will not receive gabapentin at any time during the study. Gabapentin will be administered in 400 mg tablets; placebo tablets will appear identical to the gabapentin tablets. Gradual increases in medication doses are used in order to minimize side effects and enhance compliance. At the start of week 1, the group receiving gabapentin will be administered at 400 mg three-times a day. This dose will be increased to 800 mg three-times a day at week 2 and increased to 1200 mg three-times a day at the start of week 3. The dose will continue at 1200 mg three-times a day for weeks 3 through 8. Dose reductions for tolerability will be made by the research psychiatrist in coordination with the research pharmacy. All patients must take a minimum of gabapentin/placebo 400 mg BID to remain in the study.

Both the active and placebo medication capsules will contain riboflavin, which will allow the clinic to verify that the study medication is being taken correctly and absorbed by the body. Urine samples obtained weekly will be examined under a UV lamp in order to observe any fluorescence signifying the consumption of the study capsules. The patient will consume approximately 100 mg of riboflavin daily.

The goal of compliance enhancement therapy is to achieve high quality supportive treatment as well as consistency between treatment groups. Treatment will be delivered in 9 individual sessions over 9 weeks. Sessions will last approximately 30 minutes and will be structured, focused on setting abstinence from benzodiazepine use as a goal, patient compliance, and current functioning. The therapist will promote a positive supportive therapeutic relationship with the treatment goal of encouraging abstinence from benzodiazepines and adherence to study visits and medication.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the ages of 18-65 who meet DSM-IV criteria for benzodiazepine abuse or dependence, and opioid dependence, and are being treated for opioid dependence with methadone.
* Individuals seeking treatment for benzodiazepine abuse or dependence.
* Individuals capable of giving informed consent and capable of complying with study procedures.
* Individuals must have current benzodiazepine use.
* Individuals must report using, benzodiazepines an average > 4 days per week over the past 28 days. The average amount of benzodiazepine used per using day must be > lorazepam 4 mg/day or its equivalent

  (1 mg lorazepam = 0.25 mg clonazepam = 0.5 mg alprazolam = 5 mg diazepam = 10 mg chlordiazepoxide)
* Women of child-bearing age will be included provided that they are not pregnant, based on the results of a blood pregnancy test done at the time of screening and agree to use a method of contraception with proven efficacy and not to become pregnant during the study.

Exclusion Criteria:

* Subjects with any current Axis I psychiatric disorder as defined by DSM-IV-TR supported by the SCID-I/P that in the investigator's judgment that are unstable or would be disrupted by study medication or by an effort to discontinue benzodiazepines. Disorders that are stable on psychotherapy or pharmacotherapy will not be exclusionary.
* Individuals with evidence of acute physiological benzodiazepine withdrawal.
* Individuals with a history of seizures during alcohol or sedative-hypnotic withdrawal.
* Individuals with a history of requiring pharmacologic detoxification from alcohol or sedative-hypnotic agents in the past year.
* Individuals meeting DSM IV criteria for current cocaine dependence as their primary substance use disorder diagnosis.
* Unstable physical disorders that might make participation hazardous such as uncontrolled hypertension and tachycardia (SBP > 150 mm Hg, DBP > 90 mm Hg, or a sitting quietly HR > 100 bpm), acute hepatitis (patients with chronic mildly elevated transaminase levels [2-3 x upper limit of normal] are acceptable) or poorly controlled diabetes. Kidney disease or impaired kidney function that would interfere with the excretion of gabapentin is exclusionary.
* Patients currently taking prescribed psychotropic medications, other than methadone or medications prescribed for pain syndromes, that would be disrupted by study medication or by an effort to discontinue benzodiazepines. Anticonvulsants prescribed for pain syndromes are exclusionary.
* Patients with a known sensitivity to gabapentin.
* Individuals who have exhibited suicidal or homicidal behavior within the past two years or have current active suicidal ideation.
* Women who are pregnant or nursing.
* Individuals physiologically dependent on any other drugs (excluding nicotine, caffeine, methadone).
* Individuals currently prescribed gabapentin.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2007-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John J Mariani, M.D, Principal Investigator — Columbia University/New York State Psychiatric Institute
Locations (1):
- Bridge Plaza Treatment and Rehabilitation Clinic, Long Island City, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mariani JJ, Malcolm RJ, Mamczur AK, Choi JC, Brady R, Nunes E, Levin FR. Pilot trial of gabapentin for the treatment of benzodiazepine abuse or dependence in methadone maintenance patients. Am J Drug Alcohol Abuse. 2016 May;42(3):333-40. doi: 10.3109/00952990.2015.1125493. Epub 2016 Mar 10. PMID 26962719

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gabapentin | Placebo
Started | 8 | 11
Completed | 5 | 7
Not Completed | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gabapentin | Placebo | Total
Number analyzed (Participants) | 8 | 11 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 11 | 19
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 6 | 8 | 14
Region of Enrollment [Number; unit: participants]
  United States | 8 | 11 | 19

OUTCOME MEASURES:

1. Primary Outcome: Mean Reduction Change in Benzodiazepine Use Per Day Based on Time Line Follow Back
Description: Comparing the mean reduction change in Benzodiazepine use per day when comparing the baseline week prior to study entry to the last week of study participation based on the Time Line Follow Back
Time Frame: data collected during 8 weeks of trial or length of participation
Population: a total of 16 participants had data available post randomization
Measure: Mean (Standard Deviation); unit: milligrams/day
Groups:
- Active Medication: gabapentin treatment 1200 mg three times daily
  Gabapentin: For the first week, one 400 mg Gabapentin capsule taken 3 times per day. For the second week, two 400 mg Gabapentin capsules taken 3 times per day. For the third week through the eighth week, three 400 mg Gabapentin capsules taken 3 times per day. For the ninth and last week, two 400 mg Gabapentin capsules taken 3 times per day for 3 days, then one 400 mg Gabapentin capsule taken 3 times per day for 4 days. Placebo study medication appears identical to active medication and is prescribed with an identical dosing schedule.
- Placebo: Placebo condition received pills identical in appearance to experimental arm.
  Gabapentin: For the first week, one 400 mg Gabapentin capsule taken 3 times per day. For the second week, two 400 mg Gabapentin capsules taken 3 times per day. For the third week through the eighth week, three 400 mg Gabapentin capsules taken 3 times per day. For the ninth and last week, two 400 mg Gabapentin capsules taken 3 times per day for 3 days, then one 400 mg Gabapentin capsule taken 3 times per day for 4 days. Placebo study medication appears identical to active medication and is prescribed with an identical dosing schedule.
Arm/Group | Active Medication | Placebo
Number analyzed (Participants) | 6 | 10
milligrams/day | 4.0 (4.0) | 2.3 (6.7)

ADVERSE EVENTS:
Time Frame: 8 weeks of study
Arm/Group | Gabapentin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/10
Other Adverse Events (participants affected / at risk) | 6/6 | 5/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gabapentin (N=6) | Placebo (N=10)
fatigue (General disorders) | 3 (3) | 2 (2)
somnalence (General disorders) | 5 (5) | 2 (2)
dizziness (General disorders) | 4 (4) | 0 (0)
other (General disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
An adequately powered double-blind trial is required to further evaluate the utility of gabapentin in treating benzodiazepine use disorder. Recruitment from more than one program is likely to be required to reach an adequate sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No